CLINICAL TRIAL: NCT00252629
Title: Inspiratory Flow Dynamics During Sleep in Gulf War Syndrome (GWS) and the Effect of Continuous Positive Airway Pressure (CPAP)
Brief Title: Sleep Disordered Breathing in Gulf War Illness and the Effect of Nasal CPAP Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCD-001-05S
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Results first posted 2014-12-11 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Apnea, Sleep; Chronic Fatigue Syndrome
Keywords: Fatigue; Functional Somatic Syndrome; Gulf War Syndrome; Sleep apnea; Upper Airway Resistance Syndrome
MeSH Terms: conditions — Sleep Apnea Syndromes; Fatigue Syndrome, Chronic; Fatigue; Persian Gulf Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Therapeutic nasal CPAP (Active Comparator): Comparing change of veterans reported outcomes before and after 3 weeks treatment of therapeutic nasal CPAP with the change on sham nasal CPAP.
  Interventions: Other: Nasal CPAP treatment during sleep
- Sham nasal CPAP (Sham Comparator): Comparing change of symptoms and veterans reported outcomes before and after treatment of 3 weeks on sham nasal CPAP with the change on therapeutic nasal CPAP
  Interventions: Other: Nasal CPAP treatment during sleep

INTERVENTIONS:
Other: Nasal CPAP treatment during sleep — After documenting sleep disordered breathing, GWS subject gets randomized to receive either a therapeutic nasal CPAP or a sham nasal CPAP treatment during sleep, GWS symptoms ( fatigue, pain, and cognitive dysfunction) were assessed by a baseline questionnaires and at 3 week period whether on sham or therapeutic CPAP. The change of symptoms in each group will be compared.

SUMMARY:
The purpose of this study is to determine any sleep disordered breathing in veterans with Gulf War Syndrome (GWS) and compare it to healthy normal asymptomatic Gulf War veterans. This study will also determine the effect of treatment with continuous positive airway pressure on veterans with Gulf War Syndrome.

1. The investigators hypothesize that sleep complaints (insomnia, un-refreshing sleep and daytime fatigue) among GWS patients are related to increased sleep fragmentation secondary to the presence of sleep disordered breathing in GWS patients.
2. The investigators hypothesize that increased collapsibility of the upper airway during sleep with the development of inspiratory flow limitation (IFL) and sleep disordered breathing causes the increased sleep fragmentation in GWS patients.
3. The investigators hypothesize that correction of IFL and sleep disordered breathing in GWS patients will result in an improvement of their sleep quality resulting in an improvement of their sleep complaints and other functional symptoms.

DETAILED DESCRIPTION:
Hypothesis 1: To demonstrate that compared to Gulf War Veterans without GWS, GWS patients have decreased total sleep and increased sleep fragmentation due to the presence of sleep disordered breathing

In order to accomplish this goal and subsequent goals, we will assemble two samples of Gulf War veterans. The first will be a sample of male GWS patients and the second will be a sample of male Gulf War veterans without GWS (Gulf War veteran control group).

All of the GWS patients will be registered in the Gulf War Veterans Registry. To avoid referral bias favoring the presence of IFL during sleep and sleep disordered breathing, we will enroll GWS patients by contacting them from the Registry and inviting them to participate. Gulf War veteran controls will be recruited in the same way and by advertisement. Prospective study participants will be screened on several self-report instruments to determine eligibility and assignment to the GWS group or to the Gulf War veteran control group.

Criteria for assignment to the GWS group are scores above the designated clinical cutpoint on each of three instruments measuring , fatigue, pain and cognitive dysfunction.

1. Fatigue during the preceding week will be assessed using the fatigue severity scale, a 10-item instrument measuring the level of disability related to fatigue (increasing disability rated 1-7).
2. Pain during the preceding week will be assessed using a pain visual analog scale (VAS; increasing pain rated 0-10 ).
3. Cognitive dysfunction during the preceding week, increasing difficulty with memory, ability to think, and ability to concentrate will be assessed by VAS (increasing cognitive dysfunction rated 0-10 ).

Conversely, criteria for assignment to the GW Veteran control group will require scores in the non-clinical range on each of those instruments. Every subject will have a full night polysomnogram.

Hypothesis 2: To demonstrate that the presence of IFL and sleep disordered breathing during sleep among GWS patients distinguishes them from Gulf War veterans without GWS

A second sleep study will be used to accomplish this second objective. Using precise methods, we will quantify the prevalence of IFL during sleep in GWS patients and in Gulf War veteran controls. Following completion, each study will be staged using Rechtschaffen and Kales criteria. From each study, 3 three minute periods of continuous NREM sleep (a total of approximately 120 breaths) will be randomly selected and analyzed for the prevalence of flow limited breaths. During the three minute periods, all of the breaths will be analyzed whether they occur during sleep or during brief (< 15 second) arousals.

Hypothesis 3: To demonstrate that relief of IFL during sleep and sleep disordered breathing will result in improvement of the functional symptoms of GWS patients

We will accomplish this utilizing a masked parallel group of sham-control and treatment trial of nasal continuous positive airway pressure (CPAP) in GWS patients. Functional symptoms ( fatigue, pain and cognitive dysfunction) will be assessed using validated, self-report questionnaires and daily ratings of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* First Gulf War veterans with and without the syndrome
* Males
* Between 32 and 52 years of age
* No history of current alcoholism nor opiate use
* No history of current active depression nor post-traumatic stress disorder (PTSD)

Exclusion Criteria:

* Females
* History of active alcoholism or opiate drug use
* History of active depression and PTSD

Ages: 32 Years to 52 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2005-11; Primary Completion 2008-10 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Amin, MD, Principal Investigator — VA Medical Center, Northport
Locations (1):
- VA Medical Center, Northport, Northport, New York, United States

REFERENCES:
- [Result] Amin MM, Gold MS, Broderick JE, Gold AR. The effect of nasal continuous positive airway pressure on the symptoms of Gulf War illness. Sleep Breath. 2011 Sep;15(3):579-87. doi: 10.1007/s11325-010-0406-8. Epub 2010 Aug 19. PMID 20717848
- [Result] Amin MM, Belisova Z, Hossain S, Gold MS, Broderick JE, Gold AR. Inspiratory airflow dynamics during sleep in veterans with Gulf War illness: a controlled study. Sleep Breath. 2011 Sep;15(3):333-9. doi: 10.1007/s11325-010-0386-8. Epub 2010 Aug 12. PMID 20703820

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 male veterans with GWI and Sleep Disordered Breathing recruited by advertisement, they were splitter into a matched two groups: 9 veterans received active nasal CPAP and 9 veterans received sham nasal CPAP.
  Additionally, we recruited asymptomatic 11 male veterans of Gulf war.
Groups:
- Therapeutic Nasal CPAP: Nine participants assigned to receive 3 weeks of treatment during sleep with therapeutic nasal CPAP.
  Using validated questionnaires, fatigue, pain, and cognitive dysfunction were assessed by self-report before and after the three weeks treatment trial.
  We compared the change of veterans reported outcomes "symptoms change" before and after 3 weeks treatment period on therapeutic nasal CPAP.
- Sham Nasal CPAP: Nine participants assigned to receive 3 weeks of treatment during sleep with sham nasal CPAP.
  Using validated questionnaires, fatigue, pain, and cognitive dysfunction were assessed by self-report before and after the three weeks treatment trial.
  We compared the change of veterans reported outcomes "symptoms change" before and after 3 weeks treatment period on sham nasal CPAP.
- Comparison of IFL During Sleep in GWS and Healthy: We recruited 18 male veterans with GWS (same group that were randomized to receive CPAP treatment) and 11 asymptomatic male veterans of the first Gulf war.
  All veterans had a polysomnography to determine the presence of sleep disordered breathing.
  We compared the prevalence of Inspiratory Flow Limitation (IFL) during supine stage 2 sleep among both groups.
Period: Overall Study
Arm/Group | Therapeutic Nasal CPAP | Sham Nasal CPAP | Comparison of IFL During Sleep in GWS and Healthy
Started | 9 | 9 | 11 (We used data from the 18 veterans with GWS in addition to the 11 control)
Completed | 8 (One participant assigned to therapeutic CPAP was excluded from the trial before starting treatment.) | 9 | 11 (We used data from the 18 veterans with GWS in addition to the 11 control)
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Therapeutic Nasal CPAP; Sham Nasal CPAP: The occurrence of the following 3 symptoms in a Gulf War veteran beginning after 8/90, lasting at least 6 months and present at the time of screening: fatigue that limits usual activity; musculoskeletal pain involving 2 or more regions of the body; and cognitive symptoms (memory, concentration, or attention difficulties). All 3 symptoms must be unexplained by any clearly defined organic illness.
- Healthy Asymptomatic Control: Eleven male veterans of first gulf war were screened for fatigue, pain and cognitive dysfunction by self report instrument.
  They all score below the clinical thershold and assigned as healthy asymptomatic
- Total: Total of all reporting groups
Arm/Group | Therapeutic Nasal CPAP | Sham Nasal CPAP | Healthy Asymptomatic Control | Total
Number analyzed (Participants) | 9 | 9 | 11 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (4.1) | 42.9 (3.1) | 41 (6.6) | 42.2 (0.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 9 | 9 | 11 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change of Fatigue Symptom
Description: Fatigue- increasing impact was rated 1-7 using the fatigue severity scale on days 1 and 7 averaged, where 1= no fatigue and 7= severe fatigue.
Time Frame: 3 weeks treatment with either therapeutic or sham CPAP
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Therapeutic Nasal CPAP: Comparing the change of fatigue complaint before and after 3 weeks treatment of therapeutic nasal CPAP
- Sham Nasal CPAP: Comparing the change of fatigue complaint before and after treatment of 3 weeks on sham nasal CPAP
Arm/Group | Therapeutic Nasal CPAP | Sham Nasal CPAP
Number analyzed (Participants) | 8 | 9
units on a scale | 2.1 (0.9) | 0.2 (1.0)
Statistical Analysis 1: Comparison: Therapeutic Nasal CPAP vs Sham Nasal CPAP; The change of fatigue complaint from baseline (before treatment) to post treatment ( after 3 weeks treatment) on either therapeutic CPAP or sham CPAP was compared with student t-test; Test type: Superiority or Other; p = 0.0002, t-test, 2 sided

2. Secondary Outcome: Change of Pain Complaint
Description: Pain- increased level were rated 0-10 by visual analogue scale, where 0= no pain and 10= severe pain.
  We compared the change of pain symptom before and after treatment of either 3 weeks on therapeutic nasal CPAP or sham nasal CPAP
Time Frame: 3 weeks of treatment on either therapeutic or sham nasal CPAP
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Therapeutic Nasal CPAP: Comparing the change of pain complaint before and after 3 weeks treatment of therapeutic nasal CPAP
- Sham Nasal CPAP: Comparing the change of pain complaint before and after treatment of 3 weeks on sham nasal CPAP
Arm/Group | Therapeutic Nasal CPAP | Sham Nasal CPAP
Number analyzed (Participants) | 8 | 9
units on a scale | 2.0 (0.9) | 0.4 (1.2)
Statistical Analysis 1: Comparison: Therapeutic Nasal CPAP vs Sham Nasal CPAP; The change of pain symptom from baseline (before treatment) to post treatment ( after 3 weeks treatment) on either therapeutic CPAP or sham CPAP was compared with student t-test; Test type: Superiority or Other; p = 0.0008, t-test, 2 sided

3. Secondary Outcome: Change of Cognitive Dysfunction
Description: Cognition dysfunction- increasing difficulty with memory, ability to think, and ability to concentrate was rated 0-10 daily by visual analogue scale, where 0 no problem and 10=severe problems.
Time Frame: 3 weeks treatment with either therapeutic or sham CPAP
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Therapeutic Nasal CPAP: Comparing the change of cognitive dysfunction ( increasing difficulty with memory, ability to think, and ability to concentrate) complaints before and after 3 weeks treatment of therapeutic nasal CPAP
- Sham Nasal CPAP: Comparing the change of cognitive dysfunction ( increasing difficulty with memory, ability to think, and ability to concentrate) complaints before and after 3 weeks treatment on sham nasal CPAP
Arm/Group | Therapeutic Nasal CPAP | Sham Nasal CPAP
Number analyzed (Participants) | 8 | 9
units on a scale | 2.0 (1.7) | 0.4 (1.0)
Statistical Analysis 1: Comparison: Therapeutic Nasal CPAP vs Sham Nasal CPAP; The change of cognitive dysfunction complaint from baseline (before treatment) to post treatment ( after 3 weeks treatment) on either therapeutic CPAP or sham CPAP was compared with student t-test; Test type: Superiority or Other; p = 0.004, t-test, 2 sided

4. Primary Outcome: The Prevalence of Inspiratory Flow Limitation (IFL) During Sleep in GWS.
Description: IFL was determined by plotting inspiratory flow against supra-glottic pressure for each breath sampled during continuous stage 2 sleep on a full night polysomnogram on both veterans with GWS and asymptomatic gulf war veterans.
  We expressed the prevalence of inspiratory flow limitations during sleep as the percentage of flow limited breath in the sample of both GWS and asymptomatic gulf was veterans.
Time Frame: On a full night polysomnogram
Measure: Mean (Standard Deviation); unit: percentage of flow limited breaths
Groups:
- GWS Male Group: A group of18 male veterans with GWS were examined. Each participant underwent full night polysomnogram while sleeping supine using a standard clinical monitoring for sleep and breathing. Inspiratory flow was measured using pneumotachograph and respiratory effort measured with supra-glottis catheter.
  Sampling of flow and effort during continuous stage 2 sleep was obtained and compared among both groups.
  Inspiratory flow was plotted against effort for each breath. IFL was defined as a 1 cm H2O or greater decrease in supraglotic pressure without a corresponding increase in airflow of at least 5 ml/second.
  The percentage of flow limited breath was calculated as the total number of flow limited breaths divided by the total breaths in all the samples.
- Asymptomatic Male Veterans of Gulf War.: A group of 11 asymptomatic male veterans of gulf war were examined. Each participant underwent full night polysomnogram while sleeping supine using a standard clinical monitoring for sleep and breathing. Inspiratory flow was measured using pneumotachograph and respiratory effort measured with supra-glottis catheter.
  Sampling of flow and effort during continuous stage 2 sleep was obtained and compared among both groups.
  Inspiratory flow was plotted against effort for each breath. IFL was defined as a 1 cm H2O or greater decrease in supraglotic pressure without a corresponding increase in airflow of at least 5 ml/second.
  The percentage of flow limited breath was calculated as the total number of flow limited breaths divided by the total breaths in all the samples.
Arm/Group | GWS Male Group | Asymptomatic Male Veterans of Gulf War.
Number analyzed (Participants) | 18 | 11
percentage of flow limited breaths | 96 (5) | 36 (25)
Statistical Analysis 1: Comparison: GWS Male Group; The p value was based on t-test; Test type: Superiority or Other; p = 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Groups:
- Therapeutic Nasal CPAP: Comparing change of veterans reported outcomes ( fatigue, pain and cognitive dysfunction) before and after 3 weeks treatment on therapeutic nasal CPAP with change of symptoms on sham nasal CPAP
- Sham Nasal CPAP: Comparing change of veterans reported outcomes ( fatigue, pain and cognitive dysfunction) before and after 3 weeks treatment on sham nasal CPAP with change of symptoms on therapeutic nasal CPAP
- Comparison of IFL During Sleep in GWS and Healthy: We recruited 11 asymptomatic male veterans of the first Gulf war. In addition to our 18 male veterans with GWS (same group that were randomized to receive CPAP treatment).
  All veterans had a polysomnography to determine the presence of sleep disordered breathing.
  We compared the prevalence of Inspiratory Flow Limitation (IFL) during supine stage 2 sleep among both groups.
Arm/Group | Therapeutic Nasal CPAP | Sham Nasal CPAP | Comparison of IFL During Sleep in GWS and Healthy
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes